CLINICAL TRIAL: NCT04829032
Title: GOODBYE HARTMANN. AFTER 100 YEARS HARTMANN'S PROCEDURE IS GOING TO BE ABANDONED?
Brief Title: GOODBYE HARTMANN TRIAL: 100 YEARS OF HARTMANN'S PROCEDURE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parma University Hospital (Other)
Collaborators: Fausto Catena (Unknown); Gennaro Perrone (Unknown)
Responsible Party: Principal Investigator, Mario Giuffrida, MD- General Surgery Resident, Parma University Hospital
Other Study IDs: 1244
Record Dates: First submitted 2021-03-22; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Emergencies; Colon Disease; Colo-rectal Cancer; Volvulus Colon; Intussusception; Diverticulitis; Foreign Bodies
MeSH Terms: conditions — Emergencies; Colonic Diseases; Colonic Neoplasms; Intussusception; Diverticulitis; Foreign Bodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hartmann's procedure: Evaluate the role of Hartmann's procedure in emergency setting for left-sided acute surgical colonic disease (perforated diverticulitis with purulent or fecal peritonitis; colon cancer perforation-obstruction; ischemic colitis; abdominal trauma).
  Interventions: Procedure: Hartmann's procedure
- Colonic resection with primary anastomosis: Evaluate the role of colonic resection with primary anastomosis in emergency setting for left-sided acute surgical colonic disease (perforated diverticulitis with purulent or fecal peritonitis; colon cancer perforation-obstruction; ischemic colitis; abdominal trauma).

INTERVENTIONS:
Procedure: Hartmann's procedure — Hartmann's procedure
  Groups: Hartmann's procedure

SUMMARY:
Hartmann's procedure was described for the first time in 1921 as an alternative to abdominoperineal resection for the treatment of upper rectal tumours.

Although Hartmann's procedure fell out of favour for rectal cancer after the introduction of restorative procedures, it remained the most common procedure in emergency setting for many years. Nowadays Hartmann's procedure is a useful procedure in selected cases e.g. severely ill patients with a high risk of anastomotic failure. However, restoring intestinal continuity for Hartmann patients is often associated with high morbidity, and about 70% will live with a permanent colostomy. Hartmann procedure' is a rapid and simple surgical technique intended to decrease perioperative morbidity and mortality. This technique is often performed by young surgeons Indeed, end colostomy may be necessary in situations where restoration of continuity is risky, either because of unfavorable local conditions or because a more definitive resection must be aborted due to hemodynamic instability. In the last decade the Hartmann's procedure has been revalued in many studies. In diverticular disease the results of DIVA arm of the LADIES trial showed that more patients in the primary anastomosis group were stoma free compared with patients in the Hartmann's procedure group. Other studies have observed no differences in major postoperative complications or postoperative mortality between patients undergoing primary anastomosis versus Hartmann's procedure.

Hartmann's procedure reversals were associated with a higher risk of serious postoperative complications than were stoma reversals after primary anastomosis with ileostomy.

Despite the growing evidence in favour of primary anastomosis and its inclusion as a valid treatment option for perforated diverticulitis or perforated sigmoid colon in recent clinical practice guidelines, some surgeons have been hesitant to undertake anastomosis in the setting of purulent or faecal contamination and continue to choose Hartmann's procedure to eliminate concerns about anastomotic leakage.

DETAILED DESCRIPTION:
Left-sided surgical acute colonic diseases (perforated diverticulitis with generalized peritonitis, colon perforation, large bowel obstruction, colon cancer perforation or obstruction, ischemic colitis, abdominal trauma) are still a life-threatening condition requiring urgent surgical intervention.

Despite several published randomized trials, showing that primary anastomosis with or without protective ileostomy is feasible and randomized trials for laparoscopic lavage with conflicting results, the Hartmann's procedure, described for the first time in 1921 as an alternative to abdominoperineal resection for the treatment of upper rectal tumours, is still performed in many hospitals worldwide. It remained the most common procedure for acute diverticulitis and colonic perforation in emergency setting for many years. Hartmann's procedure is safe for severely ill patients; however, restoring intestinal continuity for such patients is often associated with high morbidity leaving a great percentage of patients with (up to 50%) with a permanent stoma.

Hartmann procedure' is a rapid and simple surgical technique intended to decrease perioperative morbidity and mortality. This technique is often performed by young surgeons Indeed, end- colostomy may be necessary in situations where restoration of continuity is risky, either because of unfavourable local conditions (Hinchey IV peritonitis) or because a more definitive resection must be aborted due to hemodynamic instability. Although anastomosis at the time of surgery is an alternative approach to Hartmann's procedure, there have been concerns about the safety of this approach.

In the last decade the Hartmann's procedure has been revalued and the results of different studies [DIVA arm of the LADIES trial; DIVERTI study; Halim et Al] showed that more patients in the primary anastomosis group were stoma free compared with patients in the Hartmann's procedure group.

Several studies have observed no differences in major postoperative complications or postoperative mortality between patients undergoing primary anastomosis versus Hartmann's procedure. Hartmann's procedure reversals were associated with a higher risk of serious postoperative complications than were stoma reversals after protected primary anastomosis. The management of colorectal cancer emergencies is challenging. WSES guidelines recommend in case of perforation resection with anastomosis, with or without ileostomy. Hartmann's procedure should be preferred to simple colostomy, since colostomy appears to be associated with longer overall hospital stay and need for multiple operations, without a reduction in perioperative morbidity in patients with colorectal cancer obstruction. Resection with primary anastomosis should be preferred for uncomplicated malignant left-sided large bowel obstruction in absence of other risk factors. Patients with high surgical risk are better managed with Hartmann's procedure Despite the growing evidence in favour of primary anastomosis and its inclusion as a valid treatment option for perforated diverticulitis or perforated sigmoid colon cancer in recent clinical practice guidelines, surgeons have been reluctant to perform anastomosis. Moreover, the postoperative course of the septic patient is unpredictable and it very hard to estimate it intraoperatively.

In the setting of purulent or fecal contamination most surgeons choose Hartmann's procedure to eliminate also legal concerns about anastomotic leakage. It's important to note that most of these procedures are performed off normal working hours when maybe best colorectal expertise is lacking for decision making regarding anastomosis.

Primary study objective:

1. To evaluate the role of Hartmann's procedure in emergency setting for left-sided colonic acute surgical disease (perforated diverticulitis with purulent or fecal peritonitis; colon cancer perforation-occlusion; ischemic colitis; abdominal trauma) and the type of surgery commonly performed in different level of care hospitals.
2. To investigate which factors contribute in the choice of Hartmann's procedure instead of colon resection with primary anastomosis (Hospital characteristics, surgeon experience, time of surgery, age of patients, comorbidities, etc ) Study design: International multicenter prospective cohort study. Study population: Adult patients with left-sided colonic acute surgical disease who need surgery in an emergency setting (perforated diverticulitis with purulent or fecal peritonitis; colon cancer perforation-occlusion; ischemic colitis; abdominal trauma).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Patients admitted in Emergency setting for left-sided colonic disease (perforated diverticulitis with purulent or fecal peritonitis; large bowel perforation-obstruction; colon cancer perforation-obstruction; ischemic colitis; abdominal trauma).
* Patients who underwent urgent or emergency surgery for left-sided colonic disease (perforated diverticulitis with purulent or fecal peritonitis; large bowel perforationobstruction; colon cancer perforation-obstruction; ischemic colitis; abdominal trauma).

Exclusion Criteria:

* Aged 17 or younger.
* Elective surgery.
* Non-surgical treatment.
* Patients with personal history of colorectal cancer treated surgically.
* Patients with stoma.
* Unstable patients who benefited of damage control procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients with left-sided colonic disease who have been operated in urgent-emergency setting between March -May 2021 will be prospectively analyzed and evaluated time of surgery, patient's characteristic, hospital's characteristics. All patients who have been operated in urgent-emergency setting for left-sided colonic disease are suitable for inclusion.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of Hartmann's procedure vs colic resection with primary anastomosis performed in 3-months in urgent or emergency setting for left-sided acute colonic diseases. | 3 months
  * Etiology: perforated diverticulitis; perforated colonic cancer; large bowel perforation- obstruction; colon cancer perforation-obstruction; colon ischemia; abdominal trauma.
  * Treatment: Hartmann's procedure, colonic resection with primary anastomosis with or without diverting stoma, stoma without colic resection.

SECONDARY OUTCOMES:
Risk factors that contribute in the choice of Hartmann's procedure instead of colon resection with primary anastomosis | 3 months
  - Hospital Characteristics: hospital type (academic, non-academic teaching, categorical, secondary hospital, tertiary hospital, level 4- trauma center); annual volume of
  emergency surgical procedures; annual volume of left-sided colonic disease; types of diagnostic and treatment modalities that are available in the hospital.
  * Surgeon experience (surgeon in training: less than 50 colorectal resections performed; less than 5 resections per year in the last 5 years; Trained surgeon: more than 50 colorectal resections performed; more than 10 resections per year in the last 5 years)
  * Time of surgery: weekdays, weekend, public holidays, night shift (day: 8am- 8pm; night: 8pm-8am)
The number of patients treated with Hartmann's procedure with a permanent stoma after one year. | 1 year
  1 year follow up to evaluate the number of patients treated with Hartmann's procedure have a permanent stoma after one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Giuffrida, Parma, Italia, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT04829032/Prot_000.pdf